CLINICAL TRIAL: NCT00957476
Title: Omega-3 Supplementation Decreases Inflammation and Fetal Obesity in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Patrick Catalano, Professor Reproductive Biology, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB06-00255; R01HD057236 (NIH)
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Inflammation; Obesity; Pregnancy; Fetal Growth
Keywords: Pregnancy; Metabolic Diseases; Obesity; Fetal adiposity; Omega-3; Inflammation; Insulin Resistance
MeSH Terms: conditions — Inflammation; Obesity; Metabolic Diseases; Insulin Resistance | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fish Oil (Active Comparator): 800mg DHA & 1200mg EPA
  Interventions: Dietary Supplement: Omega-3 Fish Oil
- Placebo (Placebo Comparator): Wheat germ oil
  Interventions: Dietary Supplement: Omega-3 Fish Oil

INTERVENTIONS:
Dietary Supplement: Omega-3 Fish Oil — 800mg DHA and 1200mg EPA or the equivalent of a placebo PO (by mouth) once a day from enrollment (prior to 16 weeks gestation) until delivery.

SUMMARY:
Randomized, double-blind placebo controlled trial of fish oil to decrease inflammation in pregnancy.

DETAILED DESCRIPTION:
In addition to the increase in obesity in adult and children, there has been a significant increase in birth weights over the last 2 decades. Based on our preliminary data, maternal pre-gravid obesity is the strongest risk factor for neonatal as well as adolescent obesity. The long-term goals of our research are to examine therapeutic strategies to decrease fetal adiposity. Obesity and pregnancy are both insulin resistant conditions associated with chronic low-grade inflammation. Therefore, we hypothesize that n-3 PUFA dietary supplements during pregnancy will act as insulin sensitizers decreasing peripheral insulin resistance and inflammation. If correct this mechanism should decrease availability of maternal nutrients to the fetus and subsequently reduce adiposity at birth. We plan a prospective randomized double blind control trial of n-3 PUFA supplementation and placebo in overweight/obese women, with a previous cesarean delivery, initiated in early pregnancy and maintained throughout pregnancy. This proposal has two specific aims. Specific aim 1 is to evaluate the effect of n-3 PUFA supplementation on maternal insulin sensitivity. Measures of maternal insulin sensitivity and lipid metabolism will be made using the ISogtt, indirect calorimetry body composition (BODPOD) and plasma lipid profile at baseline and after dietary intervention.

Specific aim 2 will assess the effect of n-3 PUFA on the inflammatory status in overweight/obese pregnant women. We hypothesize that n-3 PUFA supplementation decreases chronic inflammation during pregnancy by preventing monocyte activation and accumulation of macrophages in WAT thus lowering systemic concentration of pro-inflammatory cytokines. We plan to characterize the longitudinal changes in circulating monocytes and plasma adipokines in order to define the inflammatory patterns in both groups over time. We will also determine the abundance and phenotype of macrophages infiltrating WAT using flow cytometry, immunohistochemistry and gene expression profiling. Furthermore, the role of PPARγ as a central target of n-3 PUFA action to regulate insulin sensitivity will be examined by characterizing the expression of PPARγ in WAT of both supplemented and control groups. Additionally, we will investigate the direct affect of n-3 PUFA on the expression of adiponectin and PPARγ regulated genes in primary cultured adipocytes.

In summary, this proposal combines both clinical and molecular methodologies in an overweight/obese subject population in order to assess the effect of n-3 PUFA on inflammation and insulin resistance. Preliminary data will also be obtained on fetal body composition in order to later address the prevention of the long term adverse effects (developmental programming) of maternal obesity in the developing fetus.

ELIGIBILITY:
Inclusion Criteria:

* BMI (wt/ht2) > or = 25 at first antenatal visit
* Gestational age at randomization between 8-16 weeks
* No medical problems such as hyperlipidemia, hypertension, or pregestational diabetes
* Between the ages of 18 and 40 years old
* Non-smokers
* No obstetrical problems such as a history of preeclampsia or gestational diabetes
* Confirmed singleton pregnancy

Exclusion Criteria:

* Major fetal anomaly
* Regular intake of fish oil supplements (defined as greater than 500 mg per week within the last four weeks). This is due to the placebo group receiving fish oil outside of the study.
* Daily use of nonsteroidal anti-inflammatory agents
* Allergy to fish or fish products, gluten intolerant (because the placebo contains wheat germ oil, which is not gluten free).
* Women who are vegetarians and do not eat any fish.
* Infants born preterm (less than 36 weeks gestation) or less than 2kg.
* Heparin use or known thrombophilia (thrombophilias include homozygous for Factor V Leiden).
* Moderate or high titer IgG anticardiolipin antibodies or prolonged activated PTT or other indication of presence of lupus anticoagulant, homozygous for prothrombin gene (G20210A) mutation, antithrombin III deficiency.
* Protein S (low levels outside of pregnancy) or Protein C deficiency.
* Hyperhomocysteinemia (due to safety concerns because n-3 may affect bleeding time).
* Hemophiliacs including von Willebrand's disease (because of safety concerns associated with the hemophilia treatment combined with the n-3 supplements).
* Planned termination of pregnancy.
* Current hypertension or current use of antihypertensive medication (including diuretics), due to increased risk of adverse pregnancy outcome.
* Pregestational diabetes due to increased risks of affecting fetal growth. We will not exclude women who develop GDM during pregnancy but consider a sub-analyses of these women depending on the number of subjects. Known maternal medical complications: cancer (including melanoma but excluding other skin cancers).
* Current hyperthyroidism if not adequately controlled.
* Renal disease with altered renal function (serum creatinine > 1.5).
* Epilepsy or other seizure disorder.
* Systemic lupus (not discoid lupus), scleroderma, polymyalgia rheumatic.
* Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes).
* Platelet or red blood cell disorder (including idiopathic thrombocytopenia purpura, a history of alloimmune thrombocytopenia in a previous offspring, significant anemia due to hemoglobinopathy but not sickle cell trait. Iron deficiency anemia will NOT be an exclusion as long as the hemoglobin is > 8 gm/dl).
* Chronic pulmonary disease (asthma of any degree of severity is NOT an exclusion).
* Structural, functional or ischemic heart disease. Neither mitral valve prolapse nor paroxysmal supraventricular tachycardia are considered exclusions.
* Known HIV positive with viral load greater than 1,000 copies/ml or CD4 count less than 350/mm3.
* Current or planned cerclage due to interference with the natural cause of delivery.
* Illicit drug or alcohol abuse during current pregnancy.
* At the time of birth, all infants will be evaluated by a pediatrician to make sure that they are healthy. Infants will be excluded from further study if they have any medical problems such as respiratory distress syndrome.
* Infants will also be excluded if they have any problems that exclude them from having estimation of body composition, for e.g. birth weight less than 2 kg.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Decreased inflammation during human pregnancy | enrollment (8-16 weeks) to delivery
  cytokine concentration in plasma, placenta and white adipose tissue

SECONDARY OUTCOMES:
Reduction of insulin resistance | enrollment (8-16 weeks) to delivery
  insulin sensitivity as estimated by OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Catalano, MD, Principal Investigator — MetroHealth Medical Center; Sylvie Hauguel-de Mouzon, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
when data analysis completed
Supporting Information: Study Protocol
Time Frame: when data analysis completed
Access Criteria: when data analysis completed

REFERENCES:
- [Derived] Calabuig-Navarro V, Puchowicz M, Glazebrook P, Haghiac M, Minium J, Catalano P, Hauguel deMouzon S, O'Tierney-Ginn P. Effect of omega-3 supplementation on placental lipid metabolism in overweight and obese women. Am J Clin Nutr. 2016 Apr;103(4):1064-72. doi: 10.3945/ajcn.115.124651. PMID 26961929
- [Derived] Berggren EK, Groh-Wargo S, Presley L, Hauguel-de Mouzon S, Catalano PM. Maternal fat, but not lean, mass is increased among overweight/obese women with excess gestational weight gain. Am J Obstet Gynecol. 2016 Jun;214(6):745.e1-5. doi: 10.1016/j.ajog.2015.12.026. Epub 2015 Dec 21. PMID 26719212
- [Derived] Haghiac M, Yang XH, Presley L, Smith S, Dettelback S, Minium J, Belury MA, Catalano PM, Hauguel-de Mouzon S. Dietary Omega-3 Fatty Acid Supplementation Reduces Inflammation in Obese Pregnant Women: A Randomized Double-Blind Controlled Clinical Trial. PLoS One. 2015 Sep 4;10(9):e0137309. doi: 10.1371/journal.pone.0137309. eCollection 2015. PMID 26340264